CLINICAL TRIAL: NCT04945928
Title: Safety and Feasibility of Surgery After Conversion Therapy for Locally Advanced and Advanced NSCLC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-013
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Neoplasm; Advanced Cancer; Locally Advanced Cancer
Keywords: Conversion Therapy; Lung Cancer; Locally Advanced and Advanced NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery after conversion therapy (Experimental): Participants with locally advanced or advanced NSCLC who received first-line treatment have been evaluated as resectable after multidisciplinary discussion involving the department of thoracic surgery, respiratory medicine, radiology and oncology.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Participants having been evaluated as operable after receiving first-line treatment (first-line chemotherapy, targeted therapy, immunotherapy, chemotherapy combined with immunotherapy, etc.) will receive surgery.

SUMMARY:
Lung cancer is one of the most common malignant tumors worldwide and the mortality ranks first in the world. In recent years, with the development of targeted therapy and immunotherapy, the overall survival of lung cancer patients has improved significantly. However, the inoperable advanced tumor remains the main reason for the poor prognosis of lung cancer. Thus, we aim to carry out this single-arm, prospective study to evaluate the safety and feasibility of surgery after conversion therapy for locally advanced and advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Previous studies have shown that selective surgery after conversion therapy is feasible and safe in locally advanced or stage IV patients, and indicates potential benefits for these patients. However, surgery after conversion therapy is difficult and has high risk of postoperative complications which requires strict operation indications and patient screening. At present, there are only relevant retrospective studies and no prospective evidence. Therefore, our team plans to carry out this single-arm prospective clinical trial to evaluate the safety and feasibility of surgery in patients with locally advanced and advanced non-small cell lung cancer after conversion therapy, so as to lay the foundation for further research and clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study with good compliance. Able to complete the observation and follow-up and have signed the informed consent;
* More than 18 years old with no limit of sex;
* Pathologically confirmed stage T4N0-3 or T1-3N2-3 NSCLC with residual tumor after first-line treatment (first-line chemotherapy, targeted therapy, immunotherapy, chemotherapy combined with immunotherapy, etc.) evaluated operable for radical resection; pathologically confirmed stage IVA NSCLC evaluated operable after first-line treatment (first-line chemotherapy, targeted therapy, immunotherapy, chemotherapy combined with immunotherapy, etc.);
* ASA score: I-III;
* Cardiopulmonary functions meet the requirements of radical operation for lung cancer with normal liver and kidney functions.

Exclusion Criteria:

* Serious heart, lung, liver and kidney dysfunction and unable to tolerate the operation;
* Neurologic, mental illness or mental disorder which is hard to control, poor compliance, unable to cooperate or describe the treatment response;
* Unable to receive radical resection;
* Need of palliative or emergency operation due to lung abscess or hemoptysis;
* Having received neoadjuvant chemoradiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
perioperative morbidity | postoperative in-hospital stay up to 30 days
  rate of perioperative complications, mainly include: pneumonia, arrhythmia, incision infection, vocal cord paralysis, trachea cannula

SECONDARY OUTCOMES:
lymph nodes counts | At operation day
  overall lymph node counts, number of stations dissected, and number of lymph nodes in each lymph node station
R0 rate | postoperative in-hospital stay up to 30 days
  R0 resection rate
operation time | At operation day
  duration of operation
blood loss | At operation day
  blood loss in the operation
operative complications | At operation day
  rate of adverse events happened in the operation
postoperative hospital stay | postoperative in-hospital stay up to 30 days
  length of postoperative hospitalization
30-day mortality | postoperative in-hospital stay up to 30 days
  30-day mortality after surgery
1-year overall survival (OS) | 1 year after surgery
  OS at 1 year after surgery
3-year overall survival (OS) | 3 year after surgery
  OS at 3 year after surgery
1-year disease-free survival (DFS) | 1 year after surgery
  DFS at 1 year after surgery
3-year disease-free survival (DFS) | 3 year after surgery
  DFS at 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: He-Cheng Li, doctor, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China